CLINICAL TRIAL: NCT02307773
Title: Does Use of Lidocaine Spray on an Endoscope Immediately Before Insertion Improve Patient Tolerance to Endoscopy? A Single Center, Case-Control Study.
Brief Title: Lidocaine Spray on an Endoscope to Improve Tolerance to Endoscopy
Status: Completed | Type: Observational
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Byung Hyo Cha, MD, President of Digestive Disease Center, Internal Medicine, Cheju Halla General Hospital
Other Study IDs: 2013-M08
Record Dates: First submitted 2014-12-01; First posted 2014-12-04 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-12

CONDITIONS: C.Medical Procedure; Digestive System; Disorder of Upper Gastrointestinal Tract; Tolerance
Keywords: Upper Gastrointestinal Endoscopy; Pharyngeal Anesthesia; Lidocaine; Belching; Retching; Tolerance
MeSH Terms: conditions — Eructation | interventions — Diagnosis-Related Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case Group: Treated with additional 2 puffs of the 10% lidocaine spray on the tip of endoscope before intubation with conventional pharyngeal anesthesia
  Interventions: Drug: Case Group
- Control Group: Treated with conventional pharyngeal anesthesia without further treatment.

INTERVENTIONS:
Drug: Case Group — Consecutively, all the participants were assigned to case group with additional 2 puffs of the 10% lidocaine spray on the tip of endoscope, same medication which was used for prior pharyngeal anesthesia, or to control group with conventional pharyngeal anesthesia without further treatment. Then we compared the primary outcome measures, such as, frequency of belching and retching of two groups.
  Other Names: Beracaine Spray
  Groups: Case Group

SUMMARY:
The investigators tested whether a new method which additional lidocaine spray on the tip of endoscope can increase the tolerance of examinee during endoscopy than conventional pharyngeal anesthesia alone.

DETAILED DESCRIPTION:
All the patients underwent upper gastrointestinal endoscopy were consecutively enrolled and assigned to case group treated with additional 2 puffs of the 10% lidocaine spray on the tip of endoscope before intubation or control group with conventional pharyngeal anesthesia without further treatment. And the investigators compared their baseline characteristics, past history, sedation or not, and frequency of retching and belching were measured during the endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All the patients who underwent upper gastrointestinal endoscopy in Endoscopy Room, Cheju Hall General Hospital.

Exclusion Criteria:

* advanced older or younger age (> 90, or < 15 years)
* comorbidities scored greater than III of American Society of Anestheiologists Physical Status Classification System (ASA) score
* history of hypersensitivity reaction to lidocaine
* he pregnant
* therapeutic or emergency endoscopy

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patients who underwent upper gastrointestinal endoscopy in Endoscopy Room 2, Digestive Disease Center, Halla General Hospital, Jeju, Korea were enrolled consecutively during Nov. 4 2013 - May 7 2014.
Sampling Method: Non-Probability Sample
Enrollment: 497 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Frequency of Belching and retching | Participants will be followed for the duration of hospital stay, expected average of 1-2 hours
  Belching was defined as release of gas from the digestive tract (mainly esophagus and stomach) through the mouth and retching was defined as reverse peristaltic movement of the stomach and esophagus without vomiting.

SECONDARY OUTCOMES:
Adverse events | Participants will be followed for the duration of hospital stay, expected average of 1-2 hours
  Events suspected as Aspiration pneumonia, methemoglobinemia

CONTACTS AND LOCATIONS:
Overall Officials: Byung Hyo Cha, M.D., Principal Investigator — Digestive Disease Center and Department of Internal Medicine, Cheju Halla General Hospital, Jeju, Korea
Locations (1):
- Digestive Disease Center and Department of Internal Medicine, Cheju Halla General Hospital, Jeju City, Jeju Special Self-Governing Province, South Korea

REFERENCES:
- [Background] Gordon MJ, Mayes GR, Meyer GW. Topical lidocaine in preendoscopic medication. Gastroenterology. 1976 Oct;71(4):564-9. PMID 782997
- [Background] Isenberg G. Topical anesthesia: to use or not to use--that is the question. Gastrointest Endosc. 2001 Jan;53(1):130-3. doi: 10.1067/mge.2001.112093. No abstract available. PMID 11154514
- [Background] Ramsay MA, Savege TM, Simpson BR, Goodwin R. Controlled sedation with alphaxalone-alphadolone. Br Med J. 1974 Jun 22;2(5920):656-9. doi: 10.1136/bmj.2.5920.656. PMID 4835444
- [Background] Lundell LR, Dent J, Bennett JR, Blum AL, Armstrong D, Galmiche JP, Johnson F, Hongo M, Richter JE, Spechler SJ, Tytgat GN, Wallin L. Endoscopic assessment of oesophagitis: clinical and functional correlates and further validation of the Los Angeles classification. Gut. 1999 Aug;45(2):172-80. doi: 10.1136/gut.45.2.172. PMID 10403727
- [Background] Lachter J, Jacobs R, Lavy A, Weisler A, Suissa A, Enat R, Eidelman S. Topical pharyngeal anesthesia for easing endoscopy: a double-blind, randomized, placebo-controlled study. Gastrointest Endosc. 1990 Jan-Feb;36(1):19-21. doi: 10.1016/s0016-5107(90)70915-7. PMID 2179038
- [Background] Leitch DG, Wicks J, el Beshir OA, Ali SA, Chaudhury BK. Topical anesthesia with 50 mg of lidocaine spray facilitates upper gastrointestinal endoscopy. Gastrointest Endosc. 1993 May-Jun;39(3):384-7. doi: 10.1016/s0016-5107(93)70110-8. PMID 8514070
- [Background] Soma Y, Saito H, Kishibe T, Takahashi T, Tanaka H, Munakata A. Evaluation of topical pharyngeal anesthesia for upper endoscopy including factors associated with patient tolerance. Gastrointest Endosc. 2001 Jan;53(1):14-8. doi: 10.1067/mge.2001.111773. PMID 11154482
- [Background] Hedenbro JL, Ekelund M, Jansson O, Lindblom A. A randomized, double-blind, placebo-controlled study to evaluate topical anaesthesia of the pharynx in upper gastrointestinal endoscopy. Endoscopy. 1992 Aug;24(6):585-7. doi: 10.1055/s-2007-1010550. PMID 1396370
- [Background] Karim A, Ahmed S, Siddiqui R, Mattana J. Methemoglobinemia complicating topical lidocaine used during endoscopic procedures. Am J Med. 2001 Aug;111(2):150-3. doi: 10.1016/s0002-9343(01)00763-x. No abstract available. PMID 11498069
- [Background] Gunaratnam NT, Vazquez-Sequeiros E, Gostout CJ, Alexander GL. Methemoglobinemia related to topical benzocaine use: is it time to reconsider the empiric use of topical anesthesia before sedated EGD? Gastrointest Endosc. 2000 Nov;52(5):692-3. doi: 10.1067/mge.2000.110078. No abstract available. PMID 11060205
- [Background] Abdallah HY, Shah SA. Methemoglobinemia induced by topical benzocaine: a warning for the endoscopist. Endoscopy. 2002 Sep;34(9):730-4. doi: 10.1055/s-2002-33450. PMID 12195332